CLINICAL TRIAL: NCT04298658
Title: The Impact of Insomnia on Pain, Physical Function, and Inflammation in HIV
Brief Title: The Impact of Insomnia on Pain in HIV
Acronym: HIPPI
Status: Completed | Type: Observational
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Burel Goodin, Associate Professor, University of Alabama at Birmingham
Other Study IDs: 300003778; 1R01HL147603-01 (NIH)
Record Dates: First submitted 2020-02-20; First posted 2020-03-06 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: HIV; Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Diagnosis; CD4 Lymphocyte Count; Viral Load

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum and plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- HIV and Insomnia: Participants will test positive for HIV and Insomnia.
  Interventions: Diagnostic Test: Structured Clinical Interview for Diagnostic and Statistical Manual of Mental Disorders-5 (DSM-5)sleep disorders-revised; Diagnostic Test: Resmed ApneaLink Air device (Resmed, San Diego, CA).; Other: Quantitative Sensory testing (QST); Diagnostic Test: Cluster of Differentiation 4 (CD4) and Viral load
- HIV Without Insomnia: Participants will test positive for HIV and test negative for Insomnia.
  Interventions: Diagnostic Test: Structured Clinical Interview for Diagnostic and Statistical Manual of Mental Disorders-5 (DSM-5)sleep disorders-revised; Diagnostic Test: Resmed ApneaLink Air device (Resmed, San Diego, CA).; Other: Quantitative Sensory testing (QST); Diagnostic Test: Cluster of Differentiation 4 (CD4) and Viral load
- Non HIV with Insomnia: Participants will test negative for HIV and test positive for Insomnia.
  Interventions: Diagnostic Test: Structured Clinical Interview for Diagnostic and Statistical Manual of Mental Disorders-5 (DSM-5)sleep disorders-revised; Diagnostic Test: Resmed ApneaLink Air device (Resmed, San Diego, CA).; Other: Quantitative Sensory testing (QST); Diagnostic Test: OraQuick Advance Rapid HIV 1/2 Swab test
- Non HIV Without Insomnia: Participants will test negative for HIV and test negative for Insomnia.
  Interventions: Diagnostic Test: Structured Clinical Interview for Diagnostic and Statistical Manual of Mental Disorders-5 (DSM-5)sleep disorders-revised; Diagnostic Test: Resmed ApneaLink Air device (Resmed, San Diego, CA).; Other: Quantitative Sensory testing (QST); Diagnostic Test: OraQuick Advance Rapid HIV 1/2 Swab test

INTERVENTIONS:
Diagnostic Test: Structured Clinical Interview for Diagnostic and Statistical Manual of Mental Disorders-5 (DSM-5)sleep disorders-revised — Structured Clinical Interview For DSM-5 Sleep Disorders-Revised (SCISD-R) - is a semi structured interview for diagnosing sleep disorders according to Diagnostic and Statistical Manual of Mental Disorders-5 (DSM-5)
  Other Names: Structured Clinical Interview For DSM-5 Sleep Disorders-Revised (SCISD-R)
Diagnostic Test: Resmed ApneaLink Air device (Resmed, San Diego, CA). — Home Sleep Test (HST) will measure airflow (i.e., nasal pressure) using a nasal cannula and oxygen saturation to identify apnea and hypopnea and calculate an apnea hypopnea index (AHI; number of apnea and hypopnea per hour).
  Other Names: Home Sleep Test
Other: Quantitative Sensory testing (QST) — All participants will undergo quantitative sensory testing for assessment of endogenous pain modulation using painful heat, mechanical, and cold stimuli in a laboratory session lasting approximately 1 hour.
Diagnostic Test: OraQuick Advance Rapid HIV 1/2 Swab test — Participants who have an HIV negative status will complete the OraQuick Advance Rapid HIV 1/2 Swab test to confirm negative status.
  Other Names: OraQuick
  Groups: Non HIV Without Insomnia; Non HIV with Insomnia
Diagnostic Test: Cluster of Differentiation 4 (CD4) and Viral load — Participants who have an HIV positive status will have blood tested for cluster of differentiation 4 (CD4) and Viral load to confirm positive status.
  Groups: HIV Without Insomnia; HIV and Insomnia

SUMMARY:
The overall objective of this application is to investigate the impact of insomnia on pain, physical functioning, and inflammation in people living with HIV. The two aims of this study to determine 1) whether insomnia promotes increased sensitivity and inflammatory reactivity to pain stimuli, and 2) if weekly fluctuations in insomnia burden drive changes in inflammation, pain severity, and physical functioning in people living with HIV. This research could help confirm insomnia as a therapeutic target for the suppression of pain and inflammation in people living with HIV.

DETAILED DESCRIPTION:
Experimental session 1 Resting Blood Pressure and Body Mass Index will be assessed. Participants who have an HIV negative status will complete the OraQuick Advance Rapid HIV 1/2 Swab test. Study staff will administer the Structured Interview for Sleep Disorders and administer the Rapid Estimation of Adult Literacy Measure-Short Form (REALM-SF) to determine health literacy. The night of Experimental Session 1 participant will be using a Resmed ApneaLink Air device (Resmed, San Diego, CA), to identify apnea and hypopnea and calculate an apnea hypopnea index.

Between Experimental Session 1 and Experimental Session 2 Sleep assessment: Sleep data will be collected by participants in their own homes using objective and subjective measures of their sleep. Participant instructions for how to collect and record their own sleep data will be provided at the end of study session 1. Participant will be provided with a watch-like device to wear on wrist for 7 consecutive days and nights. This watch measures physical activity and sleep.

Experimental Session 2 Resting Blood Pressure and temperature will be assessed. A sample of urine will be taken to test for illicit substances that might affect the study's results. Experimental session 2 will take place in the Center for Clinical and Translational Science (CCTS) Clinical Research Unit (CRU). A clinical Research Unit (CRU) nurse will place an intravenous (IV) cannula (small plastic tube) in the arm using a needle to draw blood at the beginning of the session and then an additional four times across the study for a total of five blood draws. Participants will complete multiple questionnaires to measure health, and experience with insomnia, pain, mood and emotions, experiences with stigma and discrimination, and how participant thinks and feels about things. All participants will undergo quantitative sensory testing for assessment of endogenous pain modulation using painful heat, mechanical, and cold stimuli in a laboratory session lasting approximately 3-4 hours. Blood will be processed and stored and then used to measure inflammation.

Weekly Follow-up Sessions Participants will then complete a battery of ecologically valid movement tasks that include: 1) Performance Battery (SPPB) which includes sitting in a chair, transitioning to a standing position, balancing tests and gait speed, and the Timed Up and Go test (TUG). A clinical Research Unit (CRU) nurse will draw a quick sample of approximately 20 milliliters from the participants arm using a butterfly needle so that CRU nurse can collect blood during the beginning of each visit.

ELIGIBILITY:
Inclusion Criteria:

HIV with Insomnia

* Confirmed HIV diagnosis
* currently a patient in the University of Alabama (UAB) 1917 HIV Clinic.
* must be currently receiving stable antiretroviral therapy (ART).
* Meets the Diagnostic and Statistical Manual of Mental Disorders-5 (DSM-5) diagnostic criteria for insomnia including sleep difficulty.

HIV Without Insomnia

* Confirmed HIV diagnosis
* currently a patient in the University of Alabama (UAB) 1917 HIV Clinic.
* must be currently receiving stable antiretroviral therapy (ART).
* Does not meet the Diagnostic and Statistical Manual of Mental Disorders-5 (DSM-5) diagnostic criteria for insomnia including sleep difficulty.

Non HIV with Insomnia

* Confirmed Non HIV diagnosis and currently not a patient in the UAB 1917 HIV Clinic.
* Meets DSM-5 diagnostic criteria for insomnia including sleep difficulty.

Non HIV Without Insomnia

* Confirmed Non HIV diagnosis and currently not a patient in the UAB 1917 HIV Clinic.
* Does not meets DSM-5 diagnostic criteria for insomnia including sleep difficulty.

Exclusion Criteria:

* concurrent medical conditions that could confound
* interpretation of sleep
* pain
* inflammatory issues or coexisting diseases
* Systemic rheumatic disease/condition
* uncontrolled hypertension (i.e., BP > 150/95)
* circulatory disorders (e.g., Reynaud's disease)
* history of heart disease or cardiac events
* history of cancer
* asthma AND use of an inhaler
* history of seizures
* history of stroke or other neurological disorder
* pregnancy
* core body temperature > 100 degrees Fahrenheit as this could indicate acute infection with fever; (k)
* unwilling to provide blood for this study
* non-English speaking
* recent injury or surgical procedure within past 6 months.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 120 individuals with HIV (60 with insomnia & 60 without insomnia) as well as a group of 120 individuals without HIV as Controls (60 with insomnia & 60 without insomnia), for a total sample size of 240 individuals.
Sampling Method: Non-Probability Sample
Enrollment: 171 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
Pro-Inflammatory markers | Baseline up to 8 weeks
  TNF-a, IL-6, IL-12, IL-18, C-reactive protein, sCD14/163, D-dimer and IFN-gamma assays will be performed on the blood to identify levels of pro-inflammatory markers.
Anti-Inflammatory markers | Baseline up to 8 weeks
  IFN-a, TGF-B, IL4, IL-10 and IL-13 assays will be performed on the blood to identify levels of anti-inflammatory markers.
Oxidative Stress markers | Baseline up to 8 weeks
  Mitochondrial DNA damage, Damage associated molecular patterns (DAMPS) and Cortisolassays will be performed on the blood to identify levels of anti-inflammatory markers.
Pain threshold | Baseline up to 1 week
  Pain threshold refers to the intensity at which a stimulus is first perceived as painful. Heat stimuli will be delivered using a computer-controlled thermal stimulation system with a 30 millimeter X 30 millimeter probe. From a baseline of 32 degrees Celsius, the probe temperature will increase at a rate of .5 degrees Celsius/second until the participant responds by pressing a button on a handheld device. For heat pain threshold, participants will be instructed to press the button when the sensation "first becomes painful"
Pain tolerance | Baseline up to 1 week
  Pain tolerance refers to the maximum amount of pain produced by a stimulus that a person is able/willing to tolerate. Heat stimuli will again be delivered using the computer-controlled thermal stimulation system. From a baseline of 32 degrees Celsius, the probe temperature will increase at a rate of .5 degrees Celsius/second until the participant responds by pressing a button on a handheld device. For heat pain tolerance, participants will be instructed to press the button when they are "no longer willing to tolerate" the painful sensation.
Punctate Stimuli | Baseline up to 1 week
  Monofilament touch test refers to the maximum amount of pain produced by a stimulus that a person is able/willing to tolerate. Participants will be asked to rate their pain after being stimulated either once or ten times with vonfrey filament, or until they can no longer tolerate" the painful sensation.
Temporal summation of pain | Baseline up to 1 week
  Temporal summation of pain refers to a form of endogenous pain facilitation characterized by the perception of increased pain despite constant or even reduced peripheral afferent input. Temporal summation is presumed to be the psychophysical manifestation of wind-up. Wind-up is a phenomenon where repetitive stimulation of C primary afferents at rates greater than 0.3 Hertz produces a slowly increasing response of second-order neurons in the spinal cord. A series of 5 heat pulses will be repeated every two seconds starting at a baseline temperature of 40 and participants will be asked to rate how painful each peak of the pulse feels to them using a pain rating of 0-100 (0 no pain at all to 100 the most intense pain imaginable). These heat pulses will be repeated randomly at three different temperatures peaking at 44, 46, and 48 degrees in Celsius.
Conditioned pain modulation | Baseline up to 1 week
  A routinely used quantitative sensory testing protocol for the measurement of endogenous pain inhibition, which refers to the reduction in pain from one stimulus (the test stimulus) produced by the application of a second pain stimulus (the conditioning stimulus). The conditioning stimulus will be the cold pressor task (Thermo Scientific) applied to the non-dominant hand. For this procedure the cold water will be maintained at 10C and participants will keep their hand immersed for 60 seconds. Upon removal of the hand, a mechanical pressure stimulus will be applied. The pressure stimulus used is a handheld, digital pressure algometer (Algomed, Medoc, Ramat Yishai, Israel) to assess pressure pain applied to the dominant forearm and ipsilateral trapezius by gradually increasing pressure at a rate of 30 kiloPascals (maximum 1000 kiloPascals) per second until participants indicate when the increasing pressure first becomes painful by pressing a button on a device they will be holding.
Actigraph Sleep Measurement | Baseline up to 8 weeks
  A light weight and compact watch-like device used for objective measurement of sleep. The device will be worn for 7 consecutive days/nights and will track physical activity, falling asleep and waking events, and includes an integrated light sensor for recording photopic light.
Weekly Sleep Diaries | Baseline up to 8 weeks
  A sleep diary including 15 daily questions will be filled out every day for seven days including questions about a participants nightly sleep experiences.
Weekly Caffeine Diaries | Baseline up to 8 weeks
  A caffeine dairy including different types of caffeine generally available for the participants to record their daily caffeine consumption of for seven days.

SECONDARY OUTCOMES:
Short Physical Performance Battery | Week 2 up to 8 weeks
  The SPPB consists of 3 individual sub-tests - standing balance (participants are asked to stand in 3 easy stances for 10 seconds), 4-meter gait speed (participants are asked to walk a steady pace in a straight line for 4-meters) and 5-repetition sit-to-stand (particpants are asked to stand up and sit back down in a stable chair up to 5 times). All 3 are simple and quick to perform in the outpatient setting and require only limited equipment; participants are asked to rate difficulty 0-100 (0 no difficulty and 100 being the most difficult imaginable) and pain 0-100 (0 no pain and 100 being the most pain imaginable).

OTHER OUTCOMES:
Timed Up and Go (TUG) Task | Week 2 up to 8 weeks
  The Timed Up and Go test (TUG) is a commonly used screening tool to assist clinicians to identify patients at risk of falling. Participants are asked to start in a sitting position in a chair, stand up and walk approximately 3 meters before turning to return to the chair at a steady, straight pace. The outcome will be measured with a stopwatch, then rating difficulty 0-100 (0 no difficulty and 100 being the most difficult imaginable) and pain 0-100 (0 no pain and 100 being the most pain imaginable).
Munich Chrono Type Questionnaires (MCTQ) | Baseline
  Consisting of 19 questions, this is a self-reported scale that is used to assess the midpoint of everyday wake and sleep schedules, as well as assessing an individual's chronotypes.
Insomnia Severity Index (ISI) | Baseline up to 8 weeks
  Using a 5-point scale and 7 questions, the ISI has each participant subjectively measure their insomnia severity.
Demographics (DEMO) | Baseline
  This questionnaire better helps the investigators understand how each participant's financial, racial, social, etc. background. It ranges from general questions such as age and birthday, to socioeconomic questions such as work status and financial stability.
Center for Epidemiological Studies - Depression (CESD) | Baseline up to 8 weeks
  By specifically asking about the past week, this questionnaire seeks to gain a better understanding of each participant's state of mind in reference to depressive behaviors and/or feelings.
RU Sated | Baseline up to 8 weeks
  Sleep is a key aspect in an individual's everyday life. This questionnaire measures overall sleep quality in six different categories---Regularity, Sleep quality, alertness, timing, efficiency, and duration. This helps investigators understand a person's sleep efficacy.
Physical Health Questionnaire (PHQ-15) | Baseline
  The main goal of this questionnaire is to assess and individual's overall health status/condition. It asks questions about a person's physical well-being, and aims to identify any illnesses they may be suffering from.
Difficulties in Emotion Regulation Scale (DERS) | Baseline
  This questionnaire aims to subjectively measure the different emotions a person may be feeling, and how difficult it may be for a person to regulate those emotions.
Dysfunctional Beliefs and Attitudes about Sleep (DBAAS) | Baseline
  This questionnaire measures various sleep related attitudes and assesses beliefs about sleep that are related to insomnia.
Pain Interference and Intensity (PI-I) | week 1 up to 7 weeks
  This questionnaire seeks to understand how pain has an influence/impacts an individual's everyday life and activities, sleep, and mood in general.
Sorge 24 Hour Food Record | Baseline up to 1 week
  Tcord provides individuals with the space to write down what they've eaten in the past 24 hours, as well as what time, where they ate it, and about how much they think that they ate.
Sorge Dietary Habits | Baseline up to 1 week
  This questionnaire asks about a person's general diet and intake.
Drug Abuse Screening Test (DAST10) | Baseline up to 1 week
  This drug screening asks questions related to the consequences of drug abuse and the problems associated with it.
State Trait Anxiety Inventory | Baseline up to 1 week
  This psychological questionnaire aims to measure the intensity of anxiety. It seeks to separate the state anxiety (temporary) from trait anxiety (general), as well as general anxiety and depressive feelings.
Penn State Cigarette Dependence Index - Cigarettes | Baseline up to 1 week
  Seeks to measure the level of addiction/dependence on smoking cigarettes.
Penn State Cigarette Dependence Index - Ecigarettes | Baseline up to 1 week
  Seeks to measure the level of addiction/dependence on smoking electronic cigarettes.
Alcohol Use Disorders Identification Test - C (AUDIT) | Baseline up to 1 week
  This questionnaire assesses alcohol consumption as well as related problems and behaviors.
Alcohol Smoking and Substance Involvement Screening Test (ASSIST) | Baseline up to 1 week
  This questionnaire detects and measures substance abuse, alcohol, and smoking as well as related problems. It aims to detect the risky behavior related to each.
Anger PROMIS | Baseline up to 1 week
  This questionnaire measures emotions, primarily anger, relevant to the past 7 days.
Perceived Stress Scale (PSS) | Baseline up to 1 week
  This 14 -item self-report scale measures the degree to which an individual perceives the amount of stress in their lives.
Pain Catastrophizing Scale (PCS) | Baseline up to 1 week
  This is a subjective look into how catastrophizing impacts an individual's pain. Specifically, it aims to measure catastrophic thinking related to pain they experience during the experimental session.
HIV Stigma Mechanisms | Baseline up to 1 week
  This questionnaire aims to see how an individual internalizes their experiences with HIV. Further, it asks about the negative feelings related and the beliefs associated with HIV.
Heightened Vigilance Scale (HVS) | Baseline up to 1 week
  Measures the different ways people anticipate experiencing discrimination in their everyday life by asking them to rate 4 items that describe how they prepare to face day to day discrimination (scale 1-6; 1 almost every day, 6 never).
Experience of Discrimination (EOD) | Baseline up to 1 week
  This scale evaluates each individual's experiences of discrimination. By providing a list of reasons a person may be discriminated against, it aims to see how each individual perceives their experiences.
Adverse Childhood Experiences (ACE) | Baseline up to 1 week
  This questionnaire scores on a 10 point scale, and asks about childhood experiences in reference to abuse and neglect.
Lee Fatigue Scale (LFS) | Baseline up to 1 week
  This 0-10 rating scale aims to assess fatigue and energy over time.

CONTACTS AND LOCATIONS:
Overall Officials: Burel R Goodin, PHd, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- UAB, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Tenorio AR, Zheng Y, Bosch RJ, Krishnan S, Rodriguez B, Hunt PW, Plants J, Seth A, Wilson CC, Deeks SG, Lederman MM, Landay AL. Soluble markers of inflammation and coagulation but not T-cell activation predict non-AIDS-defining morbid events during suppressive antiretroviral treatment. J Infect Dis. 2014 Oct 15;210(8):1248-59. doi: 10.1093/infdis/jiu254. Epub 2014 May 1. PMID 24795473
- [Background] Goodin BR, Owens MA, Yessick LR, Rainey RL, Okunbor JI, White DM, Mushatt KA, Harmon OA, Heath SL, Merlin JS. Detectable Viral Load May Be Associated with Increased Pain Sensitivity in Persons Living with HIV: Preliminary Findings. Pain Med. 2017 Dec 1;18(12):2289-2295. doi: 10.1093/pm/pnx057. PMID 28398572
- [Background] Merlin JS, Westfall AO, Heath SL, Goodin BR, Stewart JC, Sorge RE, Younger J. Brief Report: IL-1beta Levels Are Associated With Chronic Multisite Pain in People Living With HIV. J Acquir Immune Defic Syndr. 2017 Aug 1;75(4):e99-e103. doi: 10.1097/QAI.0000000000001377. PMID 28328552